CLINICAL TRIAL: NCT02830945
Title: Innovative Multigenerational Household Intervention to Reduce Stroke and CVD
Acronym: FITSMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington State University (Other)
Responsible Party: Principal Investigator, Dedra Buchwald, Principal Investigator, Washington State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01HL122148 (NIH)
Record Dates: First submitted 2016-05-24; First posted 2016-07-13 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Stroke; Cardiovascular Disease
MeSH Terms: conditions — Stroke; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Brochure Arm (Other): Control Arm households receive a culturally tailored Stroke and CVD brochure for prevention.
  Interventions: Other: Control Brochure Arm
- Motivational Interviewing Intervention Arm (Experimental): The MI intervention households receive three aspects of the intervention: digital stories, motivational interviewing talking circle and the option to receive text messages to adhere to the action plan.
  Interventions: Behavioral: Motivational Interviewing Intervention Arm

INTERVENTIONS:
Behavioral: Motivational Interviewing Intervention Arm
  Arms: Motivational Interviewing Intervention Arm
Other: Control Brochure Arm
  Arms: Control Brochure Arm

SUMMARY:
American Indians (AI's) are experiencing an epidemic of stroke morbidity and mortality, with higher prevalence and incidence, younger age at onset, and poorer survival than other racial and ethnic groups. With a stroke incidence more than twice that of the general U.S. population, stroke in AI's is a public health problem of staggering scope. AI's also have disproportionate burdens of many risk factors for stroke, including hypertension, smoking, obesity, and diabetes. However, no rigorous, population-based studies of stroke prevention have included AI's. The investigators at WSU, and community partners, have designed the "Family Intervention in the Spirit of Motivational Interviewing" (FITSMI), a program delivered at the household level to encourage lifestyle changes that transform the home environment and reduce stroke risk for all residents. FITSMI uses a "talking circle" format in which facilitators guide participants to identify goals for change and create a tailored plan for sustainable implementation that may target smoking, exercise, diet, or medication adherence. FITSMI requires just 2 sessions (baseline and 1 month post-baseline), with text messaging used to boost long-term adherence. In a group-randomized trial design, the investigators will recruit 360 households where Strong Heart Family Study members aged 45 and older reside. The investigators will assign half to FITSMI and half to a control condition that receives educational brochures.

ELIGIBILITY:
Inclusion Criteria:

* Household must include one member over the age of 45 (index participant)

Exclusion Criteria:

* Under the age of 11

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 458 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Stroke Risk Classification | 1 year
  Investigators will use the Stroke Risk Scorecard, developed by the National Stroke Association to classify the stroke risk of participants. The factors used to classify stroke risk will be collected using a questionnaire to assess the prevalence of high blood pressure, atrial fibrillation, smoking, high cholesterol, physical activity, weight, and family history of stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Lonnie Nelson, PhD, Principal Investigator — WSU-IREACH
Locations (4):
- United States (4):
  - Medstar Health Research, Phoenix, Arizona
  - Oklahoma University Health Science Center, Oklahoma City, Oklahoma
  - Missouri Breaks Industries Research Inc., Eagle Butte, South Dakota
  - Washington State University, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No